CLINICAL TRIAL: NCT02908776
Title: Gut Flora Modulation for The Prevention of Pci-Related Myocardial Injury - A Randomized, Placebo Controlled, Double Blind, Investigator-Initiated, Single Centre, Preliminary Study
Brief Title: MYocardial DAmage AND MIcrobiota STUDY
Acronym: MYDA-MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Filippo Neri General Hospital (Other)
Collaborators: MENDES S.A., Lugano, Switzerland (Unknown); Università degli studi di Bologna, Italy (Unknown)
Responsible Party: Principal Investigator, Christian Pristipino, MD, San Filippo Neri General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: v216/6/2014
Record Dates: First submitted 2016-02-09; First posted 2016-09-21 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Chronic Stable Angina; Periprocedural Myocardial Damage
MeSH Terms: conditions — Angina, Stable | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary supplement - Probiotics (Experimental): 4 sachets of Ecoviesel (probiotics) per day for at least 2 weeks before undergoing a coronary angiography with possible ad hoc angioplasty; and 2 sachets of probiotic per day after angioplasty, if performed.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Sachets with inactive substance indistinguishable from Ecoviesel
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Sachets with Streptococcus thermophilus DSM 32245: 70 billion, bifidobacteria (Bifidobacterium lactis DSM 32246, Bifidobacterium lactis DSM 32247) 40 billion, lactobacilli (Lactobacillus acidophilus DSM 32241, Lactobacillus helveticus DSM 29575, Lactobacillus paracasei DSM 32243, Lactobacillus plantarum DSM 32244, Lactobacillus brevis DSM 27961): 90 billion.
  Other Names: Ecoviesel
  Arms: Dietary supplement - Probiotics
Other: Placebo — Sachets of maltose, flavors and sylicium dioxide, indistinguishable from ecoviesel sachets.
  Arms: Placebo

SUMMARY:
MYDA-MI study is a randomized, placebo controlled, double blind study performed in San Filippo Neri Hospital, Roma, Italy. The planned study duration is 18 months. The objectives are to assess the effects of pre-treatment with probiotic Ecoviesel on the incidence and magnitude of peri-procedural myocardial damage caused by coronary angioplasty in stable patients. 250 patients with chronic stable angina scheduled for a coronary angiography and possible ad hoc angioplasty will be randomized to receive pre-treatment with Ecoviesel sachets (each sachet contains 200 billions bacteria) or Placebo. The pre-treatment dosage will be 4 sachets of probiotic Ecoviesel or placebo for at least 2 weeks before the planned procedure. In patients undergoing angioplasty the same treatment will be continued for 4 weeks after PCI with secondary outcome measures performed at the end of this second stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic stable angina scheduled for coronary angiography and possible ad hoc percutaneous coronary intervention

Exclusion Criteria:

* Age >75 y.o
* Diabetes requiring treatment
* Abnormal c-TnI level before angiography
* Immunodeficiency status
* Need for oral vitamin K antagonists
* Need for antibiotics
* Use of antibiotics or probiotics within 4 weeks of enrollment
* Cancer and diseases affecting 1 year prognosis
* Participation in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of abnormal c-TnI levels in patients undergoing coronary intervention | within 24 hours from coronary angioplasty
  Percentage of patients with plasma c-TnI>99th percentile of normality at least one blood sample among those drawn at 6, 12 a 24 h post-procedure

SECONDARY OUTCOMES:
peak of c-TnI levels in patients undergoing coronary intervention | within 24 hours from coronary angioplasty
  peak plasma c-TnI concentration in blood samples drawn at 6, 12 a 24 h post-procedure
incidence of contrast-induced renal dysfunction in all patients | within 24 hours from coronary angioplasty
  Percentage of patients with plasma creatinine>25% from baseline in least one blood sample among those drawn at 6, 12 a 24 h post-procedure
in-hospital incidence of major adverse cardiac events in patients undergoing coronary intervention | up to 30 days
  Percentage of patients with in-hospital acute myocardial infarction, death or unplanned revascularisation
changes in hs-CRP in all patients after treatment phases | within 30 days of the invasive procedure
  Change in plasma hs-CRP concentration at any visit
urine metabolomics in all patients after treatment phases | up to 30 days of the invasive procedure
  Change in urine metabolomics at any visit

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pristipino, MD, Principal Investigator — San Filippo Neri General Hospital
Locations (1):
- San Filippo Neri General Hospital, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided